CLINICAL TRIAL: NCT03466918
Title: Safety and Effectiveness of Edwards Lifesciences SAPIEN 3 Transcatheter Heart Valve (THV) in the Chinese Population
Brief Title: China S3: Safety and Effectiveness of Edwards Lifesciences SAPIEN 3 THV in the Chinese Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-08
Record Dates: First submitted 2018-02-22; First posted 2018-03-15 (Actual); Results first posted 2020-07-15 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-08

CONDITIONS: Aortic Stenosis; Symptomatic Aortic Stenosis; Aortic Regurgitation
Keywords: TAVI; TAVR; CHINA; SAPIEN 3; High Risk; Transcatheter aortic valve implantation; Transcatheter aortic valve replacement
MeSH Terms: conditions — Aortic Valve Stenosis; Aortic Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Patients with SAPIEN 3 THV (Experimental): Patients will be treated with Edwards SAPIEN 3 Transcatheter Heart Valve and Commander delivery system
  Interventions: Device: SAPIEN 3 THV with the Commander delivery system

INTERVENTIONS:
Device: SAPIEN 3 THV with the Commander delivery system — Edwards SAPIEN 3 Transcatheter Heart Valve is implanted using the Commander delivery system

SUMMARY:
To evaluate the safety and effectiveness of the SAPIEN 3 (Edwards Lifesciences, Irvine, California) transcatheter heart valve implantation (TAVI) in Chinese patients with symptomatic severe calcific aortic stenosis who are considered at high risk for surgical valve replacement.

DETAILED DESCRIPTION:
Edwards SAPIEN 3 Transcatheter Heart Valve and Commander delivery system will be used for this study.

A maximum of 60 patients with symptomatic severe calcific aortic stenosis requiring transcatheter aortic valve implantation (TAVI), who are considered high risk for surgical valve replacement who received a SAPIEN 3 THV.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who are considered to be operable and high risk for surgical valve replacement: STS Score ≥ 8 and ≤ 15 or Logistic EuroSCORE ≥ 15 and ≤ 40. If STS score is below 8 and Logistic EuroSCORE is below 15, patients should have other clinical or anatomical risk factors that would be considered high risk for surgery and documented by the heart team.
2. Severe symptomatic aortic stenosis requiring aortic valve replacement characterized by one or more of the following within 60 days prior to the index procedure: AVA < 0.8 cm2, Indexed AVA <0.5 cm2/m2, mean gradient > 40mmHg, or peak aortic jet velocity > 4.0m/sec.
3. NYHA Functional Class II or greater.
4. The study patient or the study patient's legal representative has been informed of the nature of the study, agrees to its provisions and has provided written informed consent as approved by the EC of the respective clinical site.
5. The study patient agrees to comply with all required postprocedure follow-up visits.

Exclusion Criteria:

1. Evidence of an acute myocardial infarction ≤ 1 month (30 days) before the intended treatment.
2. Aortic valve is a congenital unicuspid or is non-calcified.
3. Aortic valve is bicuspid and the patient is less than 60 years old, or the aortic valve is bicuspid with no raphe (Sievers classification type 0).
4. Anomalous coronary artery that would interfere with proper placement of the valve.
5. Mixed aortic valve disease (aortic stenosis and aortic regurgitation with predominant aortic regurgitation >3+).

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2018-05-23 (Actual); Primary Completion 2019-07-03 (Actual); Study Completion 2024-06-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Prof Junbo GE, Principal Investigator — Zhongshan Hospital and Fudan University
Locations (4):
- China (4):
  - Fuwai Hospital, CAMS&PUMC, Beijing
  - WestChina Hospital, Sichuan University, Chengdu
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou
  - Zhongshan Hospital Fudan University, Shanghai

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Each study site was allowed up to two roll-in patients. Per the protocol, roll-in patients completed all study visits and procedures but were not part of the analysis. Eight of the 58 patients enrolled were roll-in patients.
Groups:
- Patients With SAPIEN 3 THV: Patients were implanted with the Edwards SAPIEN 3 Transcatheter Heart Valve using the Commander delivery system.
Period: Overall Study
Arm/Group | Patients With SAPIEN 3 THV
Started | 58
Analysis Population (8/58 patients were roll-in patients. Roll-in patients were not included in the analysis.) | 50
Completed | 58 (All 58 patients completed the 30-day primary endpoint.)
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Patients With SAPIEN 3 THV
Number analyzed (Participants) | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 76.8 (6.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 27
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Chinese | 50
Region of Enrollment [Count of Participants; unit: Participants]
  China | 50
STS Score [Mean (Standard Deviation); unit: units on a scale] — The Society of Thoracic Surgeons (STS) Score measures patient risk of mortality or morbidity at the time of cardiovascular surgery on a scale that ranges from 0% to 100%, with higher numbers indicating greater risk.
  units on a scale | 6.0 (2.77)
NYHA Class Grouped [Count of Participants; unit: Participants] — New York Heart Association (NYHA), functional classification of heart failure based on how much a patient is limited during physical activity. The rating ranges from I-IV. I = no limitations of physical activity; II = slight limitations of physical activity, ordinary physical activity results in fatigue, palpitation, shortness of breath; III = marked limitations of physical activity, less than ordinary activity causes fatigue, palpitation, or shortness of breath; IV = unable to carry on any physical activity without discomfort, symptoms of heart failure at rest.
  Participants
    Class I/II | 9
    Class III/IV | 41

OUTCOME MEASURES:

1. Primary Outcome: All-cause Mortality
Description: All of the deaths that occurred in this population regardless of the cause.
Time Frame: 30-days
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With SAPIEN 3 THV
Number analyzed (Participants) | 50
Participants | 0

2. Secondary Outcome: Cardiovascular Mortality
Description: All of the deaths that occurred in this population due to a cardiovascular issue.
Time Frame: 30-days
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With SAPIEN 3 THV
Number analyzed (Participants) | 50
Participants | 0

3. Secondary Outcome: Non-Cardiovascular Mortality
Description: All of the deaths that occurred in this population due to a non-cardiovascular issue.
Time Frame: 30-days
Measure: Count of Participants; unit: Participants
Groups:
- Patients With SAPIEN 3 THV: Patients will be implanted with the Edwards SAPIEN 3 Transcatheter Heart Valve using the Commander delivery system.
Arm/Group | Patients With SAPIEN 3 THV
Number analyzed (Participants) | 50
Participants | 0

4. Secondary Outcome: Number of Participants With a Stroke
Description: Total number of participates with a stroke.
Time Frame: 30-days
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With SAPIEN 3 THV
Number analyzed (Participants) | 50
Participants | 1

ADVERSE EVENTS:
Time Frame: 30-days
Description: All Adverse Events are site-reported.
Arm/Group | Patients With SAPIEN 3 THV
All-Cause Mortality (participants affected / at risk) | 0/50
Serious Adverse Events (participants affected / at risk) | 13/50
Other Adverse Events (participants affected / at risk) | 48/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients With SAPIEN 3 THV (N=50)
Cardiac arrest (Cardiac disorders) | 2 (2)
Atrioventricular block complete (Cardiac disorders) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 1 (1)
Coronary artery occlusion (Cardiac disorders) | 1 (1)
Ventricular flutter (Cardiac disorders) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) — The patient presented with fracture of the left femoral neck and head within 30-days post procedure, not related to the TAVR procedure.
Vascular access site occlusion (Injury, poisoning and procedural complications) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1)
Platelet count decreased (Investigations) | 1 (2)
Dizziness (Nervous system disorders) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients With SAPIEN 3 THV (N=50)
Fibrin D dimer increased (Investigations) | 17 (17)
Troponin T increased (Investigations) | 16 (16)
Troponin increased (Investigations) | 9 (9)
Blood glucose increased (Investigations) | 3 (3)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 12 (12)
Vascular access site haemorrhage (Injury, poisoning and procedural complications) | 8 (9)
Post procedural fever (Injury, poisoning and procedural complications) | 7 (7)
Post procedural constipation (Injury, poisoning and procedural complications) | 3 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 13 (13)
Anaemia (Blood and lymphatic system disorders) | 4 (4)
Leukocytosis (Blood and lymphatic system disorders) | 3 (3)
Bundle branch block left (Cardiac disorders) | 7 (7)
Atrial fibrillation (Cardiac disorders) | 4 (4)
Atrioventricular block first degree (Cardiac disorders) | 3 (3)
Pyrexia (General disorders) | 6 (6)
Oedema peripheral (General disorders) | 4 (4)
Constipation (Gastrointestinal disorders) | 4 (4)
Ecchymosis (Skin and subcutaneous tissue disorders) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Haematuria (Renal and urinary disorders) | 3 (3)
Lung infection (Infections and infestations) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Without the Sponsor's prior written consent, the Principal Investigator shall not publish the clinical study results or any documents containing any Study information at any academic conferences or in any publications of any nature.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-22): https://cdn.clinicaltrials.gov/large-docs/18/NCT03466918/Prot_SAP_000.pdf